CLINICAL TRIAL: NCT06734897
Title: Impact of Music Therapy on Speech Intelligibility in Noise With Cochlear Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armina Kreuzer (Other)
Responsible Party: Sponsor-Investigator, Armina Kreuzer, Dr. tech., Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Musiktherapie_Erwachsene
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: Music Therapy After Cochlear Implantation
Keywords: Music therapy; rehabilitation after Cochlear Implantation; Cochlear Implant; Speech Perception in Noise

STUDY DESIGN:
Intervention Model Description: This is a randomized study with a "start group A" and a "delayed group" B. Group A will begin six months of music therapy immediately after cochlear implantation, group B six months later. Another group consists of persons who do not receive any music therapy, will form the control group. The speech intelligibility values resulting from the OLSA sentence test are compared between the three groups after six and twelve months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A will begin six months of music therapy immediately after cochlear implantation.
  Interventions: Other: music therapy after Cochlear Implantation
- Group B (Experimental): Group B is the delayed group and will start music therapy six months after group A.
  Interventions: Other: music therapy after Cochlear Implantation
- Group C (Experimental): Group C won't receive any music therapy and serves as a control group.
  Interventions: Other: no music therapy after Cochlear Implantation

INTERVENTIONS:
Other: music therapy after Cochlear Implantation — The music therapy is specially designed for the rehabilitation of CI-patients. It focuses on learning to distinguish different sound sources, especially when they occur at the same time. Training involves familiarization with different aspects of music such as rhythm, melody, and pitch while at the same time also getting to know the sound of different musical instruments, including singing. The training is also aimed at learning to concentrate on spoken instructions while the music is going on. This latter aim is fundamental to the goal of this study and plays a central role in the therapy.
  Arms: Group A; Group B
Other: no music therapy after Cochlear Implantation — Group C consists of persons who do not receive any music therapy after Cochlear Implantation.
  Arms: Group C

SUMMARY:
The aim of this clinical study is to investigate whether six months of music therapy immediately after CI implantation helps to improve speech intelligibility in noise. To investigate the effect of music therapy, a randomized study will be conducted with a "start group A" and a "delayed group" B (control group 1). Group A will start six months of music therapy immediately after cochlear implantation, group B six months later. A further control group 2 will not receive any music therapy. The speech intelligibility values resulting from the OLSA sentence test will be compared between the three groups after six and twelve months.

DETAILED DESCRIPTION:
Improved speech perception is a main objective for any hearing rehabilitation using hearing devices. Even more challenging is speech comprehension in noisy environments.

Music therapy is one of the approaches that can assist users with achieving better performance in situations of difficult listening comprehension such as speech perception in noisy environments. One such music therapy concept developed in Heidelberg is based on the parallelism of language and music, whereby targeted training using musical parameters such as rhythm, pitch and timbre can have an impact on the ability to perceive speech. At present, the fact that music therapy can help improve speech intelligibility is primarily based on research with normal hearing listeners.

Nowadays, cochlear implant technology has the primary goal to restore functional hearing and speech perception in people with bilateral severe-to-profound sensorineural hearing loss. Good results will be achieved by post lingually deafened CI users regarding the understanding of open-set sentences presented in quiet. But our surroundings are rarely quiet. Therefore, the goal of good rehabilitation must be to ensure that CI users also can cope well in our noisy environment. Music therapy is thus intended to be the crucial piece in the puzzle that enables such understanding in noisy situations.

This study aims to investigate the benefits of music therapy for cochlear implant users in terms of their speech intelligibility performance in noise. This is an explorative study to determine suitable parameters such as the time point of starting the music.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged between 18-85 years
2. Patients who undergo a new CI Implantation
3. Patients who speak German as their main language

Exclusion Criteria:

1. Patients with congenital deafness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Speech recognition threshold (SRT50) six month after Cochlear Implantation | six month after Cochlear Implantation
  The variable of primary interest is the speech recognition threshold (SRT50), measured in dB SNR (Signal-to-Noise Ratio), which leads to 50% speech understanding, as obtained using the OLSA-test following six months of music therapy immediately after implantation.

SECONDARY OUTCOMES:
values of SRT50 of group A and B at twelve months | twelve months
  The question should be clarified as to whether the two groups A and B demonstrate the same improvement after 1 year. The values of the SRT50 of both groups will be compared at twelve months. The results could provide information on whether it makes a difference whether therapy is started immediately after the operation or only after six months.
Values of SRT50 of all groups at 12 months | 12 months
  It is also of interest whether the values of the SRT50 at twelve months of group C are really significantly different compared to A and B. This will give us an overview regarding the general benefits of music therapy for speech intelligibility in noise for CI users.
subjective improvements of speech intelligibilty | 6 and 12 months
  Subjective improvements in speech intelligibility after music therapy is determined using the HISQUI (Hearing Implant Sound Quality Index) questionnaire. This is a validated questionnaire consisting of 19 items scored on a 7-point Likert scale, for quantifying the self-perceived level of auditory benefit that cochlear implant users experience in everyday listening situations. A total of between 19 and 133 points can be achieved, and, depending on the result, 5 subjective sound quality categories are determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucerne Cantonal Hospital, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
This is GCP compliant.

REFERENCES:
- [Background] Digeser F, Hast A, Hessel H, Hoppe U (2008): Einfluss von Obertönen auf die Frequenzdiskrimination bei Cochlear Implant Trägern
- [Background] Wagener KC, Kühnel V, Kollmeier B (1999b) Entwicklung und Evaluation eines Satztests für die deutsche Sprache III: Evaluation des Oldenburger Sprachtests. Z Audiol 38:86-95.
- [Background] Wagener KC, Kühnel V, Kollmeier B (1999a) Entwicklung und Evaluation eines Satztests für die deutsche Sprache I: Design des Oldenburger Satztests. Z Audiol 38:4-15.
- [Background] Schuppert M, Munte TF, Wieringa BM, Altenmuller E. Receptive amusia: evidence for cross-hemispheric neural networks underlying music processing strategies. Brain. 2000 Mar;123 Pt 3:546-59. doi: 10.1093/brain/123.3.546. PMID 10686177
- [Background] Schauwecker N, Patro A, Holder JT, Bennett ML, Perkins E, Moberly AC. Cochlear Implant Qualification in Noise Versus Quiet: Do Patients Demonstrate Similar Postoperative Benefits? Otolaryngol Head Neck Surg. 2024 May;170(5):1411-1420. doi: 10.1002/ohn.677. Epub 2024 Feb 14. PMID 38353294
- [Background] Parbery-Clark A, Strait DL, Anderson S, Hittner E, Kraus N. Musical experience and the aging auditory system: implications for cognitive abilities and hearing speech in noise. PLoS One. 2011 May 11;6(5):e18082. doi: 10.1371/journal.pone.0018082. PMID 21589653
- [Background] Patel AD. Why would Musical Training Benefit the Neural Encoding of Speech? The OPERA Hypothesis. Front Psychol. 2011 Jun 29;2:142. doi: 10.3389/fpsyg.2011.00142. eCollection 2011. PMID 21747773
- [Background] Petersen B, Mortensen MV, Gjedde A, Vuust P. Reestablishing speech understanding through musical ear training after cochlear implantation: a study of the potential cortical plasticity in the brain. Ann N Y Acad Sci. 2009 Jul;1169:437-40. doi: 10.1111/j.1749-6632.2009.04796.x. PMID 19673820
- [Background] Mirza S, Douglas SA, Lindsey P, Hildreth T, Hawthorne M. Appreciation of music in adult patients with cochlear implants: a patient questionnaire. Cochlear Implants Int. 2003 Jun;4(2):85-95. doi: 10.1179/cim.2003.4.2.85. PMID 18792140
- [Background] McDermott HJ. Music perception with cochlear implants: a review. Trends Amplif. 2004;8(2):49-82. doi: 10.1177/108471380400800203. PMID 15497033
- [Background] Looi V, Gfeller K, Driscoll V. MUSIC APPRECIATION AND TRAINING FOR COCHLEAR IMPLANT RECIPIENTS: A REVIEW. Semin Hear. 2012 Nov 1;33(4):307-334. doi: 10.1055/s-0032-1329222. Epub 2012 Nov 19. PMID 23459244
- [Background] Lima JP, Iervolino SMS, Schochat E. Musical and temporal auditory skills in cochlear implant users after music therapy. Codas. 2018 Nov 12;30(6):e20180006. doi: 10.1590/2317-1782/20182018006. English, Portuguese. PMID 30462748
- [Background] Hutter E, Grapp M, Argstatter H. [Music therapy in adults with cochlear implants : Effects on music perception and subjective sound quality]. HNO. 2016 Dec;64(12):880-890. doi: 10.1007/s00106-016-0279-7. German. PMID 27837214
- [Background] Hey M, Bohnke B, Mewes A, Munder P, Mauger SJ, Hocke T. Speech comprehension across multiple CI processor generations: Scene dependent signal processing. Laryngoscope Investig Otolaryngol. 2021 Jun 15;6(4):807-815. doi: 10.1002/lio2.564. eCollection 2021 Aug. PMID 34401506
- [Background] Haumann S, Muhler R, Ziese M, von Specht H. [Discrimination of musical pitch with cochlear implants]. HNO. 2007 Aug;55(8):613-9. doi: 10.1007/s00106-006-1485-5. German. PMID 17136415
- [Background] Gfeller K, Woodworth G, Robin DA, Witt S, Knutson JF. Perception of rhythmic and sequential pitch patterns by normally hearing adults and adult cochlear implant users. Ear Hear. 1997 Jun;18(3):252-60. doi: 10.1097/00003446-199706000-00008. PMID 9201460
- [Background] Dincer D'Alessandro H, Boyle PJ, Portanova G, Mancini P. Music perception and speech intelligibility in noise performance by Italian-speaking cochlear implant users. Eur Arch Otorhinolaryngol. 2022 Aug;279(8):3821-3829. doi: 10.1007/s00405-021-07103-x. Epub 2021 Oct 1. PMID 34596714
- [Background] Amann E, Anderson I. Development and validation of a questionnaire for hearing implant users to self-assess their auditory abilities in everyday communication situations: the Hearing Implant Sound Quality Index (HISQUI19). Acta Otolaryngol. 2014 Sep;134(9):915-23. doi: 10.3109/00016489.2014.909604. Epub 2014 Jun 30. PMID 24975453
- See also: PMID: 24975453 — https://pubmed.ncbi.nlm.nih.gov/24975453/
- See also: PMID: 34596714 — https://pubmed.ncbi.nlm.nih.gov/34596714/
- See also: PMID: 9201460 — https://pubmed.ncbi.nlm.nih.gov/9201460/
- See also: DOI:10.1007/s00106-006-1485-5 — https://www.researchgate.net/publication/225155860_Diskrimination_musikalischer_Tonhohen_bei_Patienten_mit_Kochleaimplantat
- See also: PMID: 34401506 — https://pmc.ncbi.nlm.nih.gov/articles/PMC8356868/
- See also: PMID: 27837214 — https://pubmed-ncbi-nlm-nih-gov.luks1.swissconsortium.ch/27837214/
- See also: PMID: 30462748 — https://pubmed.ncbi.nlm.nih.gov/30462748/
- See also: PMID: 23459244 — https://pubmed-ncbi-nlm-nih-gov.luks1.swissconsortium.ch/23459244/
- See also: PMID: 15497033 — https://pubmed.ncbi.nlm.nih.gov/15497033/
- See also: PMID: 18792140 — https://pubmed.ncbi.nlm.nih.gov/18792140/
- See also: PMID: 19673820 — https://pubmed.ncbi.nlm.nih.gov/19673820/
- See also: PMID: 21747773 — https://pubmed.ncbi.nlm.nih.gov/21747773/
- See also: PMID: 21589653 — https://pubmed.ncbi.nlm.nih.gov/21589653/
- See also: PMID: 38353294 — https://pubmed.ncbi.nlm.nih.gov/38353294/
- See also: PMID: 10686177 — https://pubmed.ncbi.nlm.nih.gov/10686177/
- See also: Google Scholar — https://scholar.google.com/scholar_lookup?journal=Z%20Audiol&title=Entwicklung%20und%20Evaluation%20eines%20Satztests%20f%C3%BCr%20die%20deutsche%20Sprache.%20I:%20Design%20des%20Oldenburger%20Satztests&author=K%20Wagener&author=V%20K%C3%BChnel&author=B%20Kollmeier&volume=38&publication_year=1999&pages=4-15&
- See also: Google Scholar — https://scholar.google.com/scholar_lookup?journal=Z%20Audiol&title=Entwicklung%20und%20Evaluation%20eines%20Satztestes%20f%C3%BCr%20die%20deutsche%20Sprache.%20III:%20Evaluation%20des%20Oldenburger%20Satztests&author=K%20Wagener&author=V%20K%C3%BChnel&author=B%20Kollmeier&volume=38&publication_year=1999&pages=86-95&
- See also: Google Scholar — https://scholar.google.com/scholar?hl=de&as_sdt=0%2C5&q=Digeser+F+Einfluss+von+Obert%C3%B6nen+auf+die+Frequenzdiskrimination+bei+Cochlear+Implant+Tr%C3%A4gern&btnG=